CLINICAL TRIAL: NCT06371339
Title: Feasibility Study of a Gamma Camera for Optimizing Dosimetry of Patients With Thyroid Disease Treated With Radioactive Iodine
Brief Title: Optimization With a Gamma Camera of the Individualized Patient Dosimetry in Radioiodine Therapy of Thyroid Diseases
Acronym: THIDOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Collaborators: Laboratoire IJCLab (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 23 VADS 03
Record Dates: First submitted 2024-04-05; First posted 2024-04-17 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Hyperthyroidism
Keywords: Hyperthyroidism; 131I treatment; Thyroid scintigraphy; Gamma camera
MeSH Terms: conditions — Hyperthyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with hyperthyroidism treated and monitored according to the standard practices. (Other)
  Interventions: Device: Additional acquisitions with the investigational gamma-camera " MoTI ".

INTERVENTIONS:
Device: Additional acquisitions with the investigational gamma-camera " MoTI ". — The gamma-camera MoTI will be used for the study to carry out 3 or 4 additional acquisitions (depending on the therapeutic indication) compared with those provided for in standard practice with a conventional gamma camera (Syngula).
  Patients will receive their treatment as usual in two stages:
  * 1/ Pre-therapy phase:
    1. Administration of a tracer dose of 131I (Day 0).
    2. Assessment of 131I uptake/fixation rate at Day 0, Day 1, Day 5.
    3. Determination of the therapeutic dose of 131I to be administered to the patient after collegial discussion.
  * 2/ Therapy phase:
    1. Administration of the therapeutic dose (Day 0).
    2. Thyroid scintigraphy within 4 hours of treatment before the patient returns home (Day 0).
  For the study, scintigraphic acquisitions will be carried out respectively using both the standard gamma camera Syngula and the gamma camera MoTI.

SUMMARY:
This is a pilot, single-center, prospective, open-label clinical investigation of a medical device (ambulatory gamma camera " MoTI " (Mobile Therapy Imager)) for patients with hyperthyroidism (Graves' disease, toxic nodule and toxic multiheteronodular goiter) for whom 131I treatment is indicated.

Its aim is to assess the feasibility of using this ambulatory gamma camera (MoTI) in the clinic in this patient population.

20 patients will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Patient with hyperthyroidism (Graves' disease, toxic nodular goiter (TNG) or toxic multi hetero nodular goiter (GMHNT)) relevant to an indication for 131I treatment.
3. Patient with no risk of iodine saturation.
4. Patient able to maintain a sitting position in an armchair for 10 minutes with chin raised and held by a "chin rest" with head in extension.
5. WHO index ≤ 1.
6. For non-menopausal patients, use of an effective contraceptive method at the start of the clinical investigation and throughout the clinical investigation, and a negative pregnancy test before administration of the tracer activity and the 131I therapeutic activity.
7. Patient signed informed consent prior to inclusion in the clinical investigation and prior to any specific procedure for the clinical investigation.
8. Patient affiliated to a social security scheme in France.

Exclusion Criteria:

1. Absence of clinical or biological hyperthyroidism.
2. Patient with a contraindication to 131I treatment.
3. Existence of one or more nodule(s) associated with hyperthyroidism at risk of malignancy according to EU-TIRADS and Bethesda criteria if cytopuncture performed.
4. Active orbithopathy associated with Graves' disease.
5. Contrast-enhanced examination performed within the two months prior to inclusion.
6. Use of iodised products for skin disinfection (Betadine) in the 4 weeks prior to inclusion.
7. Treatment with Amiodarone and derivatives in the 18 months prior to inclusion. (Ioduria test to rule out iodine saturation).
8. Pregnant or breast-feeding woman.
9. Patient planning pregnancy within 6 months of 131I treatment.
10. Any psychological, family, geographical or sociological condition that makes it impossible to comply with the medical monitoring and/or procedures set out in the clinical investigation protocol.
11. Any co-existing medical condition which, in the opinion of the investigator, could constitute a risk by participating in this study.
12. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
The clinical feasibility of using an ambulatory gamma camera. | Maximum 1 month for each patient.
  Clinical feasibility will be assessed according to the following dimensions:
  1. Tolerability and acceptability of the gamma camera by the patient, assessed on a Likert scale between 1 (Not tolerated) and 5 (No discomfort) - (use of a "Patient Evaluation Questionnaire").
  2. The quality of the images for the expected clinical use, assessed on a Likert scale from 1 (Not interpretable) to 5 (Totally Interpretable).
  Success is defined as a patient for whom the tolerability and image production dimensions are >=3 for both examinations (Day 0 and Day 1 of the pre-therapy phase). A failure is defined as a patient presenting with at least one criterion <3 for one of the two examinations.

SECONDARY OUTCOMES:
The level of acceptance of the gamma camera by operators for carrying out examinations | Maximum 1 month for each patient.
  The level will be assessed according to different dimensions: ergonomics, ease of handling, ease of installation, carrying out the examination and processing the examination. For each dimension, a Likert scale between 1 and 5 will be used (using a "Caregiver Evaluation Questionnaire").
The quality of the images for the expected clinical use | Maximum 1 month for each patient.
  The quality will be assessed using a Likert scale from 1 (Not Interpretable) to 5 (Fully Interpretable).
The ability of the gamma camera to generate images compatible with the Picture Archiving and Communication System (PACS) | Maximum 1 month for each patient.
  It will be assessed using a Likert scale of 1 (Totally incompatible) and 5 (Totally compatible).
The quality of the images obtained with the ambulatory gamma camera compared with those obtained during the standard examination (i.e. gamma camera used in the department, Syngula) | Maximum 1 month for each patient.
  The quality will be assessed using a Likert scale between 1 (Not at all satisfactory) and 5 (Very satisfactory).
The 131I fixation rates will be measured in percent at different times. | Maximum 1 month for each patient.

CONTACTS AND LOCATIONS:
Locations (1):
- IUCT-O, Toulouse, France